CLINICAL TRIAL: NCT04693312
Title: Injection of Dorsal Scapular n at Different Levels, Dose it Make Difference?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dorsal scapular entrapment
Record Dates: First submitted 2020-11-13; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): scalene muscle level injection of depomedrol
  Interventions: Drug: Depo medrol
- Group II (Experimental): Rheumboid muscle level injection of depomedrol
  Interventions: Drug: Depo medrol

INTERVENTIONS:
Drug: Depo medrol — local injection

SUMMARY:
Dorsal scapular nerve (DSN) entrapment syndrome is an under-recognized cause of neck and shoulder pain. DSN injuries can be the origin of a well-defined chronic pain syndrome, often referred to as DSN syndrome. DSN syndrome is often characterized by a dull ache along the medial border of the scapula.

DETAILED DESCRIPTION:
Dorsal scapular nerve syndrome typically presents with a weakness of the levator scapulae and the rhomboid muscles, and results in a winged scapula. A winged scapula is where the scapula protrudes from the patient's back and can affect the ability to lift objects or pull and push. The winging of the scapula seen with dorsal scapular nerve syndrome is not as severe as seen as injury or paralysis of the serratus anterior muscle.

Dorsal scapular nerve entrapment is a very under-recognized cause of neck and shoulder pain. The scapular winging may be subtle, and the symptoms are easily mistaken for other problems. A careful history and physical exam, along with a high index of suspicion, are necessary for accurate diagnosis and therefore appropriate treatment. Injection of the dorsal scapular nerve under ultrasound guidance can be diagnostic as well as therapeutic.

ELIGIBILITY:
Inclusion Criteria:

* scapular pain

Exclusion Criteria:

* cervical radiculopathy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
scapular pain | 3 months
  visual analog scale 1-10

SECONDARY OUTCOMES:
movement pain | 3 months
  visual analog scale 1-10
fatigue | 3 months
  disability fatigue score

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — assistant professor
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No